CLINICAL TRIAL: NCT01675089
Title: A Prospective and Randomized Trial of Zoledronic Acid to Prevent Bone Loss in the First Year After Kidney Transplantation
Brief Title: Zoledronic Acid to Prevent Bone Loss After Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0776/11; 2011/22962-3 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2012-08-23; First posted 2012-08-29 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2013-03

CONDITIONS: Renal Osteodystrophy
Keywords: bone disease; kidney transplantation; bisphosphonates
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder; Bone Diseases | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zoledronic acid (Experimental): Intravenous administration of zoledronic acid (5 mg) in a single dose at the time of kidney transplantation and vitamin D replacement.
  Interventions: Drug: Zoledronic acid
- Control (No Intervention): The control group will receive only vitamin D replacement. The aim of vitamin D replacement will be serum levels of 25 (OH) vitamin D above 30 ng/ml.

INTERVENTIONS:
Drug: Zoledronic acid — The treatment group will receive 15-minute intravenous administration of zoledronic acid (5 mg) in a single dose at the time of kidney transplantation and vitamin D replacement. The aim of vitamin D replacement will be serum levels of 25 (OH) vitamin D above 30 ng/ml.
  Other Names: Aclasta
  Arms: Zoledronic acid

SUMMARY:
The purpose of this study is to determine whether zolendronic acid, a third generation bisphosphonate, is effective in preventing bone loss in the first year after kidney transplantation.

DETAILED DESCRIPTION:
For the treatment of osteoporosis in the general population, a number of drugs reduce BMD (bone mineral density) loss and the rate of incident fractures. For instance, bisphosphonates improve BMD, reduce hip fracture rates and decrease mortality in post-menopausal women. Because of lack of data on safety and an increased risk of adverse effects, the use of these drugs is controversial in patients with chronic kidney disease (CKD) and abnormalities of PTH or vitamin D, an estimated glomerular filtration rate (GFR) less than 30 ml/min/1.73m² (CKD stages 4 and 5) and after transplantation. The efficacy of short and long term bisphosphonate treatment after kidney transplantation has been examined; however, histomorphometric and fracture rate reduction data are lacking.

The purpose of this study is to determine whether zolendronic acid, a third generation bisphosphonate, is effective in preventing bone loss in the first year after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* All adult kidney transplant recipients who were stable perioperative and able to return for regular follow-up

Exclusion Criteria:

* Glomerular filtration rate < 30 ml/min/1.73m² one week after transplantation
* Previous parathyroidectomy or diagnosis of adynamic bone disease (with bone biopsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Differences in bone turnover | 1 year
  Bone histomorphometric data will be analyzed at baseline and after 1 year of kidney transplantation.

SECONDARY OUTCOMES:
Bone microarchitecture | 1 year
  Bone microarchitecture will be examined by high-resolution peripheral quantitative computed tomography at the time of transplant and after 12 months.
Changes in Bone Mineral Density | 1 year
  Bone mineral density (BMD) measurements by dual-energy X-ray absorptiometry (DEXA) will be made at the time of transplant and after 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Elias David-Neto, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clinicas - Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil